CLINICAL TRIAL: NCT02231593
Title: Pilot Testing of SAGIT in Patients With Acromegaly in Clinical Practice
Brief Title: SAGIT for Classification of Patients With Acromegaly in Clinical Practice
Acronym: SAGIT Pilot
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-52030-257
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acromegalic patients
  Interventions: Other: SAGIT

INTERVENTIONS:
Other: SAGIT — SAGIT is a Clinician-Reported Outcomes (ClinROs) tool

SUMMARY:
The purpose of this pilot study is to test SAGIT (Signs and symptoms - Associated comorbidities - GH concentration level - IGF-1 - Tumour). SAGIT is a Clinician-Reported Outcomes (ClinROs) tool developed to describe patients with acromegaly. This study will determine the potential use of a finalised operational version for patient classification in clinical practice and studies.

In addition, this study intends to carry out a qualitative evaluation of the acceptability of SAGIT by the practicing endocrinologist in terms of relevance, ease of use, applicability and usefulness of the tool in practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years-old or above
* Patient with diagnosis of acromegaly with the presence of pituitary adenoma, elevated IGF-1 and lack of serum GH suppression after oral glucose tolerance test (OGTT)
* Controlled/stable, active and treatment naïve patients.
* Patient with the cognitive and linguistic capacities to understand the information letter of the study
* Patient who signed informed consent

Exclusion Criteria:

* History of non-compliance or inability to reliably receive treatment in the foreseeable future
* Gaps in treatment of greater than 1 month within the 12 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acromegaly patients registered with endocrinologists (hospital-based or outpatient clinics)
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of acromegaly patients classified using SAGIT | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (21):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - NW Pituitary Center and Neurological Surgery, Portland, Oregon
- Brazil (4):
  - Federal University of Minas Gerais, Belo Horizonte
  - Private practice, Curitiba
  - Private practice, Saúde
  - University of São Paulo Medical School, São Paulo
- France (3):
  - CHU Bicetre, Le Kremlin-Bicêtre
  - Hôpital Huriez, CHRU DE Lille, Lille
  - CHU Rennes Hôpital sud, Rennes
- Germany (3):
  - Praxisgemeinschaft an der Kaisereiche, Wilhelm-Hauff-Straße 21, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - LMU München, München
- Italy (4):
  - Azienda Ospedaliera Spedali Civil di Brescia, Brescia
  - Montichiari Hospital, Montichiari
  - Azienda Ospedaliera Città della Salute e della Scienza, Torino
  - San Giovanni Battista Hospital, Torino
- Spain (2):
  - Hospital Universitario La Coruna, A Coruña
  - Universitary Hospital Virgen de la Vitoria, Málaga
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Leeds General Infirmary, Leeds
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Giustina A, Bevan JS, Bronstein MD, Casanueva FF, Chanson P, Petersenn S, Thanh XM, Sert C, Houchard A, Guillemin I, Melmed S; SAGIT Investigator Group. SAGIT(R): clinician-reported outcome instrument for managing acromegaly in clinical practice--development and results from a pilot study. Pituitary. 2016 Feb;19(1):39-49. doi: 10.1007/s11102-015-0681-2. PMID 26377024